CLINICAL TRIAL: NCT02867709
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo Controlled Single Attack Study to Evaluate the Efficacy, Safety, and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine
Brief Title: Efficacy, Safety, and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine
Acronym: ACHIEVE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBR-MD-02
Record Dates: First submitted 2016-08-12; First posted 2016-08-16 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Migraine, With or Without Aura
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ubrogepant 25 mg (Experimental): 1 ubrogepant 25 milligram (mg) tablet, orally for treatment of a qualifying migraine attack. Participants had the option to take a second dose, placebo-matching ubrogepant tablet or rescue medication, orally, 2 to 48 hours after initial dose.
  Interventions: Drug: Ubrogepant; Drug: Placebo-matching Ubrogepant
- Ubrogepant 50 mg (Experimental): 1 ubrogepant 50 mg tablet, orally for treatment of a qualifying migraine attack. Participants had the option to take a second dose, placebo-matching ubrogepant tablet or rescue medication, orally, 2 to 48 hours after initial dose.
  Interventions: Drug: Ubrogepant; Drug: Placebo-matching Ubrogepant
- Placebo (Placebo Comparator): 1 placebo-matching ubrogepant tablet, orally for treatment of a qualifying migraine attack. Participants had the option to take placebo-matching ubrogepant tablet or rescue medication, orally, 2 to 48 hours after initial dose.
  Interventions: Drug: Placebo-matching Ubrogepant

INTERVENTIONS:
Drug: Ubrogepant — Ubrogepant tablet(s) orally for the treatment of a qualifying migraine attack.
  Arms: Ubrogepant 25 mg; Ubrogepant 50 mg
Drug: Placebo-matching Ubrogepant — Placebo-matching ubrogepant tablet(s) orally for the treatment of a qualifying migraine attack.

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of 2 doses of ubrogepant (25 and 50 mg) compared to placebo for the acute treatment of a single migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd edition, beta version
* Migraine onset before age 50
* History of migraines typically lasting between 4 and 72 hours if untreated or treated unsuccessfully and migraine episodes are separated by at least 48 hours of headache pain freedom
* History of 2 to 8 migraine attacks per month with moderate to severe headache pain in each of the previous 3 months.

Exclusion Criteria:

* Difficulty distinguishing migraine headache from tension-type other headaches
* Has taken medication for acute treatment of headache (including acetaminophen, nonsteroidal anti-inflammatory drugs [NSAIDs], triptans, ergotamine, opioids, or combination analgesics) on 10 or more days per month in the previous 3 months
* Has a history of migraine aura with diplopia or impairment of level of consciousness, hemiplegic migraine, or retinal migraine
* Has a current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy
* Required hospital treatment of a migraine attack 3 or more times in the previous 6 months
* Has a chronic non-headache pain condition requiring daily pain medication
* Has a history of malignancy in the prior 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Has a history of any prior gastrointestinal conditions (eg, diarrhoea syndromes, inflammatory bowel disease) that may affect the absorption or metabolism of investigational product; participants with prior gastric bariatric interventions which have been reversed are not excluded
* Has a history of hepatitis within previous 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1686 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adele Thorpe, Study Director — Allergan
Locations (109):
- United States (109):
  - Clinical Research Advantage, Inc./Simon Williamson Clinic, Birmingham, Alabama
  - Clinical Research Advantage, Inc./East Valley Family Physicians, PLC, Chandler, Arizona
  - St. Joseph's Hospital & Medical Center - Barrow Neurologic Institute (BNI), Phoenix, Arizona
  - Clinical Research Advantage, Inc./Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Mayo Clinic Arizona, May Clinic Scottsdale, Scottsdale, Arizona
  - Radiant Research Inc., Tucson, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Axiom Research, LLC, Apple Valley, California
  - Hope Clinical Research, Canoga Park, California
  - Axiom Research, LLC, Colton, California
  - Pharmacology Research Institute, Encino, California
  - Neuro-Pain Medical Center, Fresno, California
  - California Headache and Balance Center, Fresno, California
  - Sun Valley Research Center, Imperial, California
  - Grossmont Center For Clinical Research, La Mesa, California
  - Pharmacology Research Institute, Los Alamitos, California
  - California Advanced Neurotherapeutic, Inc., Los Angeles, California
  - Cedars Sinai Pain Center, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Desert Valley Research, Rancho Mirage, California
  - George J Rederich MD, Inc, Redondo Beach, California
  - Artemis Institute For Clinical Research, San Diego, California
  - Clinical Research Advantage, Inc./Cassidy Medical Group-Vista, Vista, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Radiant Clinical Research, Washington D.C., District of Columbia
  - Aventura Neurological Associates, Aventura, Florida
  - Clinical Research South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Broward Research Group, Hollywood, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Neurology Associates, P.A., Maitland, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - QPS MRA, LLC (Miami Research Associates), South Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - The Kaufmann Clinic, Inc., Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Clinical Research Advantage, Inc./Michigan Avenue Internists, Chicago, Illinois
  - Cedar Crosse Research Center, Chicago, Illinois
  - Robbins Headache Clinic, Riverwoods, Illinois
  - Josephson Wallack Munshower Neurology P.C., Indianapolis, Indiana
  - Norton Neurology Services MS Services, Louisville, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Seton Medical Group, Baltimore, Maryland
  - Overlea Personal Physicians, Baltimore, Maryland
  - BTC of New Bedford, New Bedford, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - New England Regional Headache Center, Inc., Worcester, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - The Headache Center, Ridgeland, Mississippi
  - Clinical Research Advantage, Inc./Prairie Fields Family Medicine, PC, Fremont, Nebraska
  - Clinical Research Advantage, Inc, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Hope Research Institute, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Princeton Medical Institute, Princeton, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - DENT Neurosciences Research Center, Amherst, New York
  - Cushing Neuroscience Institute North Shore-LIJ Medical Group, Great Neck, New York
  - ProHealth Care Associates, LLP, Plainview, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Westchester Neuro. Const, Yonkers, New York
  - Carolina Headache Institute, Durham, North Carolina
  - Headache Wellness Center, PC, Greensboro, North Carolina
  - Lake Shore Clinical Research, LLC, Mooresville, North Carolina
  - Raleigh Neurology Associates, PA, Raleigh, North Carolina
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Radiant Research, Inc., Akron, Ohio
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - University of Cincinnati Dept of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Abington Neurological Associates, Ltd., Willow Grove, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Vista Clinical Research, Columbia, South Carolina
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Middle Tennessee Clinical Research, Fayetteville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Baptist Memorial Medical Group (Neurology Specialist - Headache Clinic), Memphis, Tennessee
  - Texas Neurology, P.A., Dallas, Texas
  - Radiant Research, Inc, Dallas, Texas
  - Research Trials Worldwide, LLC, Humble, Texas
  - Advanced Research Institute, Ogden, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - iNeuro Headache Specialist, McLean, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Blue Ridge Research Center, LLC, Roanoke, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Summit Research Network Seattle, LLC, Seattle, Washington
  - South Puget Sound Neurology, Tacoma, Washington
  - West Virginia University, Department of Neurology, Morgantown, West Virginia
  - Medical College of Wisconsin, Department of Neurology, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105
- [Derived] Johnston KM, Powell L, Popoff E, Harris L, Croop R, Coric V, L'Italien G. Rimegepant, Ubrogepant, and Lasmiditan in the Acute Treatment of Migraine Examining the Benefit-Risk Profile Using Number Needed to Treat/Harm. Clin J Pain. 2022 Nov 1;38(11):680-685. doi: 10.1097/AJP.0000000000001072. PMID 36125279
- [Derived] Lipton RB, Singh RBH, Revicki DA, Zhao S, Shewale AR, Lateiner JE, Dodick DW. Functionality, satisfaction, and global impression of change with ubrogepant for the acute treatment of migraine in triptan insufficient responders: a post hoc analysis of the ACHIEVE I and ACHIEVE II randomized trials. J Headache Pain. 2022 Apr 25;23(1):50. doi: 10.1186/s10194-022-01419-7. PMID 35468729
- [Derived] Blumenfeld AM, Knievel K, Manack Adams A, Severt L, Butler M, Lai H, Dodick DW. Ubrogepant Is Safe and Efficacious in Participants Taking Concomitant Preventive Medication for Migraine: A Pooled Analysis of Phase 3 Trials. Adv Ther. 2022 Jan;39(1):692-705. doi: 10.1007/s12325-021-01923-3. Epub 2021 Dec 7. PMID 34874514
- [Derived] Hutchinson S, Silberstein SD, Blumenfeld AM, Lipton RB, Lu K, Yu SY, Severt L. Safety and efficacy of ubrogepant in participants with major cardiovascular risk factors in two single-attack phase 3 randomized trials: ACHIEVE I and II. Cephalalgia. 2021 Aug;41(9):979-990. doi: 10.1177/03331024211000311. Epub 2021 Apr 19. PMID 33874756
- [Derived] Hutchinson S, Dodick DW, Treppendahl C, Bennett NL, Yu SY, Guo H, Trugman JM. Ubrogepant for the Acute Treatment of Migraine: Pooled Efficacy, Safety, and Tolerability From the ACHIEVE I and ACHIEVE II Phase 3 Randomized Trials. Neurol Ther. 2021 Jun;10(1):235-249. doi: 10.1007/s40120-021-00234-7. Epub 2021 Feb 20. PMID 33608814
- [Derived] Goadsby PJ, Blumenfeld AM, Lipton RB, Dodick DW, Kalidas K, M Adams A, Jakate A, Liu C, Szegedi A, Trugman JM. Time course of efficacy of ubrogepant for the acute treatment of migraine: Clinical implications. Cephalalgia. 2021 Apr;41(5):546-560. doi: 10.1177/0333102420970523. Epub 2020 Nov 26. PMID 33241721
- [Derived] Lipton RB, Dodick DW, Ailani J, Lu K, Finnegan M, Szegedi A, Trugman JM. Effect of Ubrogepant vs Placebo on Pain and the Most Bothersome Associated Symptom in the Acute Treatment of Migraine: The ACHIEVE II Randomized Clinical Trial. JAMA. 2019 Nov 19;322(19):1887-1898. doi: 10.1001/jama.2019.16711. PMID 31742631
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Started | 563 | 561 | 562
Safety Population: Received Study Drug | 499 | 478 | 488
Completed | 493 | 474 | 487
Not Completed | 70 | 87 | 75
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Withdrawal of Consent | 7 | 9 | 8
Not completed — Lost to Follow-up | 17 | 20 | 20
Not completed — Lack of Qualifying Event | 42 | 55 | 42
Not completed — Protocol Violation | 3 | 2 | 3
Period: Safety Follow-up Period
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Started | 493 | 474 | 487
Completed | 482 | 459 | 473
Not Completed | 11 | 15 | 14
Not completed — Withdrawal of Consent | 1 | 8 | 6
Not completed — Lost to Follow-up | 10 | 5 | 7
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Ubrogepant 25 mg: 1 ubrogepant 25 mg tablet, orally for treatment of a qualifying migraine attack. Participants had the option to take a second dose, placebo-matching ubrogepant tablet or rescue medication, orally, 2 to 48 hours after initial dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg | Total
Number analyzed (Participants) | 563 | 561 | 562 | 1686
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.2) | 41.6 (12.3) | 41.0 (12.4) | 41.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 501 | 497 | 1492
  Male | 69 | 60 | 65 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 449 | 467 | 456 | 1372
  Black or African American | 94 | 82 | 93 | 269
  Asian | 8 | 6 | 5 | 19
  American Indian or Alaska Native | 4 | 1 | 4 | 9
  Native Hawaiian/Other Pacific Islander | 1 | 1 | 1 | 3
  Multiple | 7 | 4 | 3 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 116 | 129 | 125 | 370
  Not Hispanic or Latino | 447 | 432 | 437 | 1316

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pain Freedom at 2 Hours After Initial Dose
Description: Pain freedom was defined as a reduction in headache pain severity from moderate/severe at baseline to no pain at 2 hours after the initial dose of investigational product. Participants were provided with electronic diary (eDiary) to rate headache severity on a scale from no pain to severe pain. Number analyzed is the number of participants with non-missing postdose pain severity assessment at or before 2 hours after initial dose.
Time Frame: Baseline (Predose) to 2 hours after initial dose
Population: Modified Intent-to-Treat (mITT) population included all randomized participants who received at least 1 dose of study drug, recorded a baseline migraine headache severity measurement, and had ≥ 1 postdose migraine headache severity or migraine-associated symptom measurement at or before the 2-hour timepoint, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 456 | 435 | 464
percentage of participants | 14.3 | 20.7 | 21.8
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.0285, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, medication use for migraine prevention, baseline headache severity were explanatory variables in model; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.09 to 2.22]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0129, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.14 to 2.29]

2. Primary Outcome: Percentage of Participants With Absence of the Most Bothersome Migraine-Associated Symptom Identified at Baseline at 2-Hours After Initial Dose
Description: The most bothersome migraine-associated symptom was the symptom (photophobia, phonophobia or nausea) present at pre-dose baseline identified by the participant to be 'most bothersome'. Participants were provided with an eDiary to record absence or presence of migraine-associated symptoms. Number analyzed is the number of participants with non-missing postdose most bothersome migraine-associated symptoms assessed.
Time Frame: Baseline (Predose) to 2 hours after initial dose
Population: mITT population included all randomized participants who received at least 1 dose of investigational product, recorded baseline migraine headache severity measurement, had ≥1 postdose migraine headache severity/migraine-associated symptom measurement at/before 2-hour timepoint, LOCF. Number analyzed is participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 456 | 434 | 463
percentage of participants | 27.4 | 34.1 | 38.9
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.0711, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, underlying symptom as explanatory variables; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.02 to 1.83]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0129, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.25 to 2.20]

3. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours After the Initial Dose
Description: Pain relief was defined as a reduction of a moderate/severe migraine headache to a mild headache or to no headache. Participants were provided with an eDiary to rate headache severity on a scale from no pain to severe pain. Number analyzed is the number of participants with non-missing pain severity assessment at or before 2 hours after initial dose.
Time Frame: Baseline (Predose) to 2 hours after initial dose
Population: mITT population included all randomized participants who received at least 1 dose of investigational product, recorded a baseline migraine headache severity measurement, and had ≥ 1 postdose migraine headache severity or migraine-associated symptom measurement at or before the 2-hour timepoint, LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 456 | 435 | 464
percentage of participants | 48.2 | 60.5 | 62.7
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.0711, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.25 to 2.17]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0129, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.35 to 2.32]

4. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 24 Hours After Initial Dose
Description: Sustained pain relief was defined as a pain relief at 2 hours with no administration of either rescue medication or the second dose of study drug, and with no occurrence thereafter of a moderate/severe headache up to 24 hours after dosing with study drug. Participants were provided with an eDiary to rate headache severity on a scale from no pain to severe pain. Determinable cases: participants for whom sustained pain relief from 2 to 24 hours status can be determined based on the observed headache severity at scheduled time points, use of rescue medication or optional second dose between 2 and 24 hours, and the answer to the headache recurrence question at 24 hours. Number analyzed is the number of participants with assessment of determinable sustained pain relief from 2 to 24 hours after initial dose.
Time Frame: 2 to 24 hours after initial dose
Population: mITT population included all randomized participants who received at least 1 dose of investigational product, recorded a baseline migraine headache severity measurement, and had ≥ 1 postdose migraine headache severity or migraine-associated symptom measurement at or before the 2-hour timepoint, determinable cases.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 443 | 424 | 449
percentage of participants | 21.0 | 32.5 | 36.7
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.0711, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.33 to 2.48]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0129, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.59 to 2.92]

5. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours After Initial Dose
Description: Sustained pain freedom was defined as a pain freedom at 2 hours with no administration of either rescue medication or the second dose of study drug, and with no occurrence thereafter of a mild/moderate/severe headache up to 24 hours after dosing with study drug. Participants were provided with an eDiary to rate headache severity on a scale from no pain to severe pain. Determinable cases: participants for whom sustained pain relief from 2 to 24 hours status can be determined based on the observed headache severity at scheduled time points, use of rescue medication or optional second dose between 2 and 24 hours, and the answer to the headache recurrence question at 24 hours. Number analyzed is the number of participants with assessment of determinable sustained pain freedom from 2 to 24 hours after initial dose.
Time Frame: 2 to 24 hours after initial dose
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 451 | 432 | 457
percentage of participants | 8.2 | 12.7 | 14.4
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.0711, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.04 to 2.53]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0129, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.20 to 2.83]

6. Secondary Outcome: Percentage of Participants With the Absence of Photophobia at 2 Hours After the Initial Dose
Description: Photophobia was defined as sensitivity to light, a migraine-associated symptom. Participants were provided with an eDiary to record absence or presence photophobia. Number analyzed is the number of participants with non-missing postdose photophobia assessment at or before 2 hours after initial dose.
Time Frame: 2 hours after initial dose
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 456 | 435 | 464
percentage of participants | 35.5 | 39.3 | 43.8
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.1833, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, photophobia were explanatory variables; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.96 to 1.72]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0167, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.14 to 2.02]

7. Secondary Outcome: Percentage of Participants With the Absence of Phonophobia at 2 Hours After the Initial Dose
Description: Phonophobia was defined as sensitivity to sound, a migraine-associated symptom. Participants were provided with an eDiary to record absence or presence of phonophobia. Number analyzed is the number of participants with non-missing postdose phonophobia assessment at or before 2 hours after initial dose.
Time Frame: 2 hours after initial dose
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 456 | 435 | 464
percentage of participants | 46.3 | 53.6 | 54.1
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.1066, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, phonophobia were explanatory variables; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.04 to 1.83]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.0440, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.05 to 1.84]

8. Secondary Outcome: Percentage of Participants With Absence of Nausea at 2 Hours After the Initial Dose
Description: Nausea was a migraine-associated symptom. Participants were provided with an eDiary to record absence or presence of nausea. Number analyzed is the number of participants with non-missing postdose nausea assessment at or before 2 hours after initial dose.
Time Frame: 2 hours after initial dose
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
Number analyzed (Participants) | 456 | 435 | 464
percentage of participants | 70.0 | 70.6 | 71.3
Statistical Analysis 1: Comparison: Placebo vs Ubrogepant 25 mg; Test type: Superiority; p = 0.9522, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; Treatment group, historical triptan response, migraine prevention medication, baseline headache severity, nausea were explanatory variables; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.81 to 1.49]
Statistical Analysis 2: Comparison: Placebo vs Ubrogepant 50 mg; Test type: Superiority; p = 0.9522, Regression, Logistic — P-value was adjusted for multiple comparisons across primary and secondary endpoints and multiple doses; [statistical method as in outcome 8, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.83 to 1.51]

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after the last dose of study drug (approximately 30 days)
Description: Safety population, all participants who received at least 1 dose of investigational product, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Placebo | Ubrogepant 25 mg | Ubrogepant 50 mg
All-Cause Mortality (participants affected / at risk) | 0/499 | 0/478 | 0/488
Serious Adverse Events (participants affected / at risk) | 0/499 | 1/478 | 0/488
Other Adverse Events (participants affected / at risk) | 0/499 | 0/478 | 0/488
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=499) | Ubrogepant 25 mg (N=478) | Ubrogepant 50 mg (N=488)
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT02867709/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT02867709/SAP_001.pdf